CLINICAL TRIAL: NCT01004224
Title: A Phase I, Open-label, Multi-center, Dose Escalation Study of Oral BGJ398, a Pan FGF-R Kinase Inhibitor, in Adult Patients With Advanced Solid Malignancies
Brief Title: A Dose Escalation Study in Adult Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398X2101; 2009-010876-73 (EudraCT Number)
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Advanced Solid Tumors With Alterations of FGFR1, 2 and or 3; Squamous Lung Cancer With FGFR1 Amplification; Bladder Cancer With FGFR3 Mutation or Fusion; Advanced Solid Tumors With FGFR1 Amplication; Advanced Solid Tumors With FGFR2 Amplication; Advanced Solid Tumors With FGFR3 Mutation
Keywords: advanced solid tumors; lung cancer; bladder cancer; BGJ398; FGFR; kinase inhibitor; advanced solid malignancies
MeSH Terms: conditions — Lung Neoplasms; Urinary Bladder Neoplasms | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BGJ398 (Experimental)
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398

SUMMARY:
The study will determine the maximum tolerated dose and thus the recommended phase II dose and schedule of the compound and characterize the safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically confirmed advanced solid tumors with FGFR1 or FGFR2 amplification or FGFR3 mutation, for which no further effective standard anticancer treatment exists
* Adequate bone marrow function
* Adequate hepatic and renal function
* Adequate cardiovascular function
* Contraception.

  * For women: Must be surgically sterile, post-menopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period; must have a negative serum or urine pregnancy test and must not be nursing.
  * For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 3 months after the treatment period

Exclusion Criteria:

* Patients with primary CNS tumor or CNS tumor involvement
* Patients with history and/or current evidence of endocrine alteration of calcium-phosphate homeostasis
* History and/or current evidence of ectopic mineralization/ calcification including but not limited to the soft tissue, kidneys, intestine, myocard and lung with the exception of calcified lymphnodes and asymptomatic coronary calcification
* Current evidence of corneal disorder/ keratopathy incl. but not limited to bullous/ band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis etc., confirmed by ophthalmologic examination.
* History or current evidence of cardiac arrhythmia and/or conduction abnormality
* Women who are pregnant or nursing.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-12-11 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate and category of dose-limiting toxicities will be tabulated for patients included in the dose escalation portion of the study, to establish the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RPTD) | 23 months
  Incidence rate and category of dose-limiting toxicities will be tabulated for patients included in the dose escalation portion of the study, to establish the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RPTD). This will be calculated using an established statistical model, based on incidence of adverse events and serious adverse events, physical examinations, vital signs, electrocardiograms, and laboratory parameters

SECONDARY OUTCOMES:
To assess preliminary anti-tumor activity of BGJ398 for patients in expansion Arm 4 (previously treated patients with advanced/metastatic UCC with FGFR3 gene alterations) | 23 months
  overall response rate (ORR), as assessed by investigator per RECIST v 1.0; overall survival (OS), duration of response (DOR) and disease control rate (DCR) will be assessed
To determine the pharmacokinetic (PK) profiles of oral BGJ398 | 23 months
  Time vs. concentration profiles, PK parameters of BGJ398 and known active metabolite(s).
To evaluate the pharmacodynamic effect of the drug. | 23 months
  Pre- vs. post treatment serial changes in FGF23 plasma levels (not done for patients enrolled to expansion Arm 4)
Assess preliminary anti-tumor activity for patients not in Arm 4. | 23 months
  Overall tumor response rate (ORR) and PFS assessed by investigator per RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (15):
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Los Angeles, California
  - University of Colorado Dept. of Anschutz Cancer (3), Aurora, Colorado
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center Onc. Dept.., New York, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital Onc Dept, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Salt Lake City, Utah
- Novartis Investigative Site, Heidelberg, Victoria, Australia
- Novartis Investigative Site, Vienna, Austria
- France (9):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Suresnes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Marburg
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Meldola, FC, Italy
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Novartis Investigative Site, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No